CLINICAL TRIAL: NCT03441438
Title: Mechanisms of Alcohol Sensitivity in Aspirin Exacerbated Respiratory Disease
Brief Title: Mechanisms of Alcohol Sensitivity in AERD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20382
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Aspirin-Sensitive Asthma With Nasal Polyps; Samter's Syndrome
Keywords: alcohol sensitivity; red wine; aerd
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Patients without asthma or aspirin intolerance who may or may not react to alcoholic beverages
  Interventions: Dietary Supplement: Water; Dietary Supplement: Red wine; Dietary Supplement: Polyphenolic Compounds
- Aspirin Tolerant Asthma (Active Comparator): Patients with asthma who are tolerant to aspirin and/or other NSAIDs and note sensitivity to alcoholic beverages
  Interventions: Dietary Supplement: Water; Dietary Supplement: Red wine; Dietary Supplement: Polyphenolic Compounds
- Aspirin Intolerant Asthma / AERD (Active Comparator): Patients with AERD who note sensitivity to alcoholic beverages
  Interventions: Dietary Supplement: Water; Dietary Supplement: Red wine; Dietary Supplement: Polyphenolic Compounds

INTERVENTIONS:
Dietary Supplement: Water — Serum and urine markers will be obtained after drinking 5 oz of water
Dietary Supplement: Red wine — Serum and urine markers will be obtained after drinking 5 oz of water
Dietary Supplement: Polyphenolic Compounds — Serum and urine markers will be obtained after consuming 100 mg of provinols powder

SUMMARY:
The purpose of this study is to determine what type of reactions in the body may be responsible for the respiratory symptoms that occur when patients with Aspirin Exacerbated Respiratory Disease (AERD) drink alcoholic beverages. These reactions are most often seen with red wine.

DETAILED DESCRIPTION:
This is a prospective trial of approximately 60 subjects with AERD to explore the mechanisms behind the physiologic reactions that occur when drinking alcoholic beverages. At various time points patients will be asked to ingest a variety of substances found in red wine after which blood and urine markers of the reaction will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Controls - must be 21 years or older
* Aspirin Tolerant Asthma and AERD arms must note a sensitivity to alcoholic beverages

Exclusion Criteria:

* Enzymopathies
* Mastocytosis
* Alcoholism
* Prior severe respiratory reaction to alcohol consumption
* Current pregnancy
* Monoamine Oxidase Inhibitor (MAOI) use
* Age under 21
* Use of leukotriene modifier 1 week before study intervention
* Having undergone and maintained aspirin desensitization

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
24 Hour Urinary Leukotriene-E4 (LTE4) | 24 hour
  Urine LTE4 ng/mg Cr

SECONDARY OUTCOMES:
24 Hour Urinary Prostaglandin-D2 (PGD2) metabolite | 24 hour collection
  Urine PGD2 metabolite ng/mg Cr
Whole blood Activated Basophil Level | 2 hours after ingestion
  Proportion of activated basophils in whole blood after ingestion
Whole Blood Activated Eosinophil Level | 2 hours after ingestion
  Proportion of activated eosinophils in whole blood after ingestion
Whole Blood tryptase | 2 hours after ingestion
  Level of tryptase concentration in whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Spencer C Payne, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Cardet JC, White AA, Barrett NA, Feldweg AM, Wickner PG, Savage J, Bhattacharyya N, Laidlaw TM. Alcohol-induced respiratory symptoms are common in patients with aspirin exacerbated respiratory disease. J Allergy Clin Immunol Pract. 2014 Mar-Apr;2(2):208-13.. doi: 10.1016/j.jaip.2013.12.003. PMID 24607050
- [Background] Payne SC. Re: Alcohol-induced respiratory symptoms are common in patients with aspirin exacerbated respiratory disease. J Allergy Clin Immunol Pract. 2014 Sep-Oct;2(5):644. doi: 10.1016/j.jaip.2014.05.003. No abstract available. PMID 25213072